CLINICAL TRIAL: NCT02338024
Title: Enhancing Linkage to HIV Care for Newly Detected HIV-positive Persons in Ukraine
Acronym: MARTAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ukrainian Institute on Public Health Policy (Other)
Responsible Party: Principal Investigator, Oleksandr Neduzhko, Researcher, Ukrainian Institute on Public Health Policy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3U01GH000752-01 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: HIV
Keywords: Enrollment in HIV care; Recently detected HIV-positive; specialized health care clinics; Ukraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MARTAS intervention (Experimental): Structured motivational sessions and further communication between linkage coordinators and HIV-positive patients focused on engagement in HIV medical care.
  Interventions: Behavioral: Modified Antiretroviral Treatment Access Study intervention
- Standard of care (No Intervention): Oral referrals to a network of government AIDS Centers or their departments ("Trust" offices) located in each study region.

INTERVENTIONS:
Behavioral: Modified Antiretroviral Treatment Access Study intervention
  Arms: MARTAS intervention

SUMMARY:
This study proposes to assess whether a modified Antiretroviral Treatment Access Study intervention, proved to be effective in the U.S. and based on the nurse case management approach, can impact the enrollment in HIV care of recently detected HIV-positive patients in specialized health care clinics in three regions in Ukraine, using the existing local infrastructure. The proposed study addresses a significant public health issue of non-/late enrollment of HIV-positive persons in HIV care and treatment.

DETAILED DESCRIPTION:
Individual, parallel, two-arm, 1:1 RCT. The study participants were recruited between October 2015 and December 2016 at 9 clinics located in Dnipropetrovsk region (Dnipropetrovsk Regional Narcological Dispensary; Dnipropetrovsk Regional Dermatovenereologic Dispensary; Kryvyi Rih Infectious Disease Clinic No. 1), Mykolaiv region (Mykolaiv Regional Narcological Dispensary; Mykolaiv Regional Dermatovenereologic Dispensary; Mykolaiv Regional Infectious Disease Clinic), and Odesa region (Odesa Regional Dermatovenereologic Dispensary; Odesa Infectious Disease Clinic; Odesa Regional Center of Mental Health). These three types of clinical sites (treating addiction, sexually transmitted infections [STIs], and infectious diseases [IDs]) were located in the regions with the highest HIV prevalence in Ukraine, but were not co-located with HIV care facilities. Participants assigned to the standard of care (SOC) arm and the MARTAS arm received referrals to the local AIDS Centers (Dnipropetrovsk Regional AIDS Center, Kryvyi Rih AIDS Center, Mykolaiv Regional Center for Palliative Care and Integrated Services (former Mykolaiv AIDS Center), and Odesa Regional AIDS Center) or their departments ("Trust" offices) located in each study region. Investigators affiliated with The Ukrainian Institute on Public Health Policy (UIPHP) were responsible for all aspects of study design, management, and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years;
* Tested HIV-positive
* Fluent in Russian or Ukrainian;
* Able to read/understand and sign an informed consent

Exclusion Criteria:

* Enrolled in HIV care;
* Plan to move out of the study region before the end of their follow-up period
* Cognitive impairment
* Have pending legal issues, independent of their lifetime history of incarceration
* Subject is a part of another intervention or/and research study with similar linkage-to-care objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
The proportion of referred intervention patients who enroll in HIV care | 3 months
  Linkage (registration) to HIV care within the 3-month period after study enrollment-both self-reported and confirmed by the medical record.

CONTACTS AND LOCATIONS:
Locations (10):
- Ukraine (10):
  - Dermatovenereological dispensary, Dnipropetrovsk
  - Narcological dispensary, Dnipropetrovsk
  - Infectious disease clinic, Kryvyi Rih
  - Ukrainian Institute on Public Health Policy, Kyiv
  - Dermatovenereological dispensary, Mykolaiv
  - Infectious disease clinic, Mykolaiv
  - Narcological dispensary, Mykolaiv
  - Center of psychical health, Odesa
  - Dermatovenereological dispensary, Odesa
  - Infectious disease clinic, Odesa

REFERENCES:
- [Derived] Neduzhko O, Postnov O, Sereda Y, Kulchynska R, Bingham T, Myers JJ, Flanigan T, Kiriazova T. Modified Antiretroviral Treatment Access Study (MARTAS): A Randomized Controlled Trial of the Efficacy of a Linkage-to-Care Intervention Among HIV-Positive Patients in Ukraine. AIDS Behav. 2020 Nov;24(11):3142-3154. doi: 10.1007/s10461-020-02873-7. PMID 32333208